CLINICAL TRIAL: NCT02174224
Title: Program Evaluation of a Hospital-based Violence Intervention Program (At-risk Intervention and Mentoring)
Brief Title: At-risk Intervention and Mentoring Evaluation
Acronym: AIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Denver Health and Hospital Authority (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: OJJDP-2013-3579
Record Dates: First submitted 2014-06-23; First posted 2014-06-25 (Estimated); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Violence
Keywords: Violence; At-risk youth; Intentional Injury; Violence Intervention; Youth; recidivism
MeSH Terms: conditions — Recidivism | interventions — Crisis Intervention; Case Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SMC + BI + Case Management (Experimental): This arm will include all interventions in Standard Medical Care + Brief Intervention Arm. Case management will also be given to this arm. General needs based assessments will be conducted by the outreach worker. These assessments will be done at the hospital or at the youth's home, whichever they prefer. This assessment tool addresses education, vocational training, employment, housing, medical insurance, follow-up care and pro-social activities. Although each youth in this arm will receive the same needs-based assessment, individual youth will have variable needs, which will guide each unique and individualized case management plan.
  Interventions: Behavioral: Brief Intervention; Behavioral: Case Management; Behavioral: Standard Medical Care

INTERVENTIONS:
Behavioral: Brief Intervention — Goals of the bedside intervention will be to help the patient understand their risky behaviors that resulted in the injury and to assess and deescalate any threat of retaliatory violence by the patient. The outreach worker will: (1) develop a rapport with the patient by introducing themselves and describing their (outreach worker's) background and reason for the bedside visit; (2) assess the emotional response to the current injury; (3) ensure the patient and/or family understand the nature of the injury and ED course; (4) address any immediate concerns of the patient; and (5) develop a plan for staying safe following discharge.
Behavioral: Case Management — Case management based on needs-assessment. Resource connection and mentoring.
Behavioral: Standard Medical Care — This will include physician discretion for medical treatment and potentially a social worker visit as the physician sees fit for the patient. This will also include a list of resources that are typically needed and used for violently injured youth.

SUMMARY:
The purpose of this study is to determine if a hospital-based violence intervention programs can make sustainable behavior changes in at-risk youth using two key components, brief intervention at the hospital bedside and case management.

DETAILED DESCRIPTION:
This study will be a randomized controlled trial. Youth presenting to the emergency department with an intentional injury (gunshot wound, stab wound, or assault) will be given a behavioral assessment. Participants will be categorized according to risk (low, moderate, high). Only moderate or high youth will continue in the study and be randomized. Low risk youths will receive the medical standard of care and be re-assessed at 18 months.

Randomization will place participants in one of two arms. Arm 1 will receive the standard of care PLUS a brief intervention with AIM outreach workers. Arm 2 will receive standard medical care PLUS a brief intervention PLUS case management.

Every randomized youth will be assessed for risk and protective factors and have have data collected at 6-month intervals (0, 6, 12, 18 months).

ELIGIBILITY:
Inclusion Criteria:

* 14-24 years of age , Intentional Injury (Gunshot Wound, Stab Wound, Assault)

Exclusion Criteria:

* Younger than 14, 25 or older, non-English speaking, unable to give informed consent/assent, sexual assaults, domestic violence, child neglect/abuse.

Ages: 14 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 133 (Actual)
Dates: Start 2014-06; Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Violence Risk Scale | 0, 6, 12, 18 months
  Violence Risk Scale (VRS) will be measured with each youth at 4 time points. Change over time will be assessed and compared among study arms.

SECONDARY OUTCOMES:
Composite Score | 0, 6, 12, 18 months
  Composite Score measures both risk and protective factors. This weighted scale uses the interplay between risk and protective factors to determine overall risk for youth to become violently injured.
School Enrollment | 0, 6, 12, 18 months
  Self-report for school enrollment will be measured and compared among arms.
Hospital Recidivism | 0, 6, 12, 18 months
  Every six month, patients' medical records will be scanned to determine if there has been violent injury recidivism. Medical release of Information forms will allow medical record searches from other local hospitals.
Justice System Recidivism | 0, 6, 12, 18 months
  Self-report of criminal history.
Employment | 0, 6, 12, 18 months
  Self-report of employment status.
Resource Utilization | 0, 6, 12, 18 months.
  Self report of resource utilization for health care and social needs.
Mortality | 0, 6, 12, 18 months
  Mortality will be assessed every 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Katie Bakes, MD, Principal Investigator — Denver Health Medical Center
Locations (1):
- Denver Health Medical Center, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No